CLINICAL TRIAL: NCT04970537
Title: Efficacy Analysis of Tigecycline-based Therapy and Polymyxin B-based Therapy in ICU Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 202105202
Record Dates: First submitted 2021-07-04; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2020-08

CONDITIONS: Tigecycline; Polymyxin B; Intensive Care Unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The gender, age, ICU diagnosis, basic diseases, antibiotic treatment plan, physiological indicators, duration of hospital stay, length of stay in ICU, hospitalization cost, prognosis and other discharge information of patients receiving tigecycline or polymyxin B admitted to the ICU of four provincial-level Grade A hospitals in Changsha, Hunan Province ,China from 2017 to 2021 were included.

To analyze the therapeutic effect of tigecycline-based or polymyxin B-based antibiotic regimens and their effect on the prognosis of patients, and to conduct subgroup analysis.

DETAILED DESCRIPTION:
The gender, age, ICU diagnosis, basic diseases, antibiotic treatment plan, physiological indicators, duration of hospital stay, length of stay in ICU, hospitalization cost, prognosis and other discharge information of patients receiving tigecycline or polymyxin B admitted to the ICU of four provincial-level Grade A hospitals in Changsha, Hunan Province ,China from 2017 to 2021 were included. The four hospitals included the 1st-3th XiangYa Hospitals and Hunan Provincial People's Hospital. Organize the data.Patients with a course of treatment < 4 days and shedding were excluded.To analyze the therapeutic effect of tigecycline-based or polymyxin B-based antibiotic regimens and their effect on the prognosis of patients, and to conduct subgroup analysis. The chi-square test was used for the counting data, and the Mann-Whitney U test or Kruskal-Wallis H test was used for the measurement data. The significance value was adjusted by Bonferroni correction method for multiple tests, and the P was tested on both sides,P>0.05.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients receiving tigecycline or polymyxin B treatment;
* Age 14-95, gender unlimited;
* there are clear infections and strains;
* The patient and/or his/her family agree to sign the informed consent voluntarily.

Exclusion Criteria:

* Patients with treatment of less than 4 days;
* patients with abscission;
* Pregnant patients;
* Patients with age < 14 years or > 95 years.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 14-95 year-old patients in ICU, who received tigecycline and polymyxin B treatment (≥4d).
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2017-07-23 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
hospital mortality rate | up to hospital discharge or die in hospital, up to 48 weeks(estimation).
  Patients die in hospital or abandon treatment due to poor prognosis in hospital after treatment of tigecycline or polymyxin B
30d mortality rate | up to the 30th day of the treatment of tigecycline or polymyxin B
  Patients die after treatment of tigecycline or polymyxin B
Bacterial clearance rate | from the first day of the treatment of tigecycline or polymyxin B until to the end day, up to 8 weeks (estimation).
  Bacterial clearance during treatment of tigecycline or polymyxin B

SECONDARY OUTCOMES:
The length of hospital stay | up to hospital discharge or die in hospital, up to 48 weeks (estimation).
  The length of hospital stay,days
The length of ICU stay | up to hospital discharge or die in hospital, up to 24 weeks (estimation).
  The length of ICU stay
Hospitalization Cost | up to hospital discharge or die in hospital, up to 48 weeks (estimation).
  total Hospitalization Cost
serum creatinine | at the end day of the treatment of tigecycline or polymyxin B, up to 8 weeks (estimation).
  serum creatinine at the end day of the treatment of tigecycline or polymyxin B
MV days | up to hospital discharge or die in hospital, up to 48 weeks (estimation).
  the total days with mechanical ventilation
VA days | up to hospital discharge or die in hospital, up to 48 weeks (estimation).
  the total days with vasoactive agent

CONTACTS AND LOCATIONS:
Overall Officials: Shuangping Zhao, Study Chair — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital of Central south university, Changsha, Hunan, China